CLINICAL TRIAL: NCT00189982
Title: Recombinant Antihemophilic Factor Manufactured and Formulated Without Added Human or Animal Proteins (ADVATE rAHF-PFM): Safety Monitoring in Pediatric Patients Diagnosed With Severe to Moderately Severe Hemophilia A - A Continuation of Baxter Clinical Study 060101
Brief Title: Efficacy and Safety Study of a Recombinant and Protein-Free Factor VIII (rAHF-PFM) in Pediatric Patients in Canada With Hemophilia A - A Continuation of Baxter Study 060101
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060401
Record Dates: First submitted 2005-09-08; First posted 2005-09-19 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
Keywords: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A

INTERVENTIONS:
Drug: Antihemophilic Factor Manufactured and Formulated without Added Human or Animal Proteins (rAHF-PFM) — Treatment regimens were determined by the investigator, and may have been any combination of standard prophylaxis (25 to 50 IU/kg body weight, 3 to 4 times per week), investigator-determined prophylaxis, and/or on-demand treatment (dose selected by investigator). Once the treatment regimen was established, the regimen was to be maintained for the duration of the study, unless clinical reasons necessitated a change.
  The treatment of bleeding episodes and perioperative management was at the discretion of the investigator and consistent with the institution's standard of care.

SUMMARY:
The purpose of this study is to evaluate whether rAHF-PFM is safe and effective in the treatment of children with hemophilia A. The study is open to pediatric patients in Canada who completed Baxter Study 060101.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have participated and completed participation in Baxter's clinical study 060101
* Subject or parent/legally authorized representative has provided written informed consent

Exclusion Criteria:

* Subjects who have withdrawn from Baxter's Clinical Study 060101 prior to the termination of the study

Max Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2004-12-17 (Actual); Primary Completion 2006-11-10 (Actual); Study Completion 2006-11-10 (Actual)

PRIMARY OUTCOMES:
Assessment of safety, as measured by the incidence, causality, and severity of adverse experiences | Throughout the study period of approximately 23 months.

SECONDARY OUTCOMES:
Assessment of the hemostatic efficacy in the treatment of bleeding episodes; | At least 50 exposure days or a total treatment time of 6 months, whichever came first.
assessment of the hemostatic efficacy in surgical or invasive procedures | From day of surgery until time of discharge from hospital or clinic (up to approximately 2 weeks post surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada